CLINICAL TRIAL: NCT04550546
Title: Effects of Nystatin Suspension Oral Application on Oral Microbial Community
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jin Xiao, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004638
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Nystatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nystatin treatment (Experimental): Participants will be given 1-week supply of nystatin suspension (6ml 600,000 U/mL) and be instructed to rinse the mouth with nystatin for 1 minute and spit out the suspension, at a frequency of four times a day, for a duration of 1 week. Participants will be instructed to spit the suspension after the oral rinse and do not swallow the suspension, and they will be instructed to avoid eating, drinking and brushing their teeth for 30 minutes.
  Interventions: Drug: Nystatin

INTERVENTIONS:
Drug: Nystatin — 600,000 U/mL of nystatin in a rinse suspension

SUMMARY:
The purpose of this study is to examine the effect of a prescription mouth rinse (Nystatin),an FDA approved drug, on the different types of bacteria in the mouth. Results from this study may help understand the effect that Nystatin oral rinse has on certain types of oral bacteria, which may also cause tooth decay.

DETAILED DESCRIPTION:
This is a prospective, single-arm clinical trial of patients diagnosed with oral candidiasis.

designed clinical study. All study participants will have positive oral Candida detection with sufficient oral Candida burden to meet the laboratory criteria for a diagnosis of oral candidiasis (≥ 400 CFU/mL of salivary Candida, a standard that was established by Dr. Epstein at the Department of Oral Diagnosis and Department of Microbiology and Immunology at the University of Washington in 1980). All study participants will receive treatment for oral candidiasis using nystatin suspension (Brand name: Mycostatin), and be instructed to rinse the mouth with (6ml of 600,000 U/mL) nystatin suspension, followed by spitting out the suspension, at the frequency of four times per day, for a period of 1 week. The oral microbial changes including fungal and cariogenic bacteria (e.g. S. mutans) will be monitored immediately (within 7 days) and 3-months following the completion of the 1-week Nystatin application. Detailed inclusion and exclusion criteria and methods see below.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in this study and able to come for follow-up appointments.
* Has positive oral Candida detection and the amount of oral Candida meet the laboratory criteria for diagnosing oral Candidiasis (>= 400 colony forming unit in saliva).
* Has ≥ 10,000 CFU/mL of S. mutans in the saliva (justification: individuals with ≥ 10,000 CFU/mL salivary S. mutans are considered at elevated risk for dental caries).
* Ability to consent, comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* visible signs of candidiasis on the mucosa or tongue at screening (Patients will be referred for treatment immediately)
* Patient with systemic diseases, such as HIV, cancer or diabetes. This will be answered by study participants and further confirmed by using electronic medical record (EPIC) for those participants who have records in the EPIC system. (Justification: patient with systemic diseases is that patients with these conditions are more prone to yeast and bacterial infection)
* History of local (oral) or systemic antibiotics or antifungal medication within the last 3 months. This will be answered by study participants and further confirmed by using electronic medical record (EPIC) for those participants who have records in the EPIC system.
* Women who are currently pregnant or reported that she is currently breast feeding . A pregnancy test (urine test) will be conducted to exclude participants who are pregnant. Rational of excluding pregnant women and women are currently breastfeeding their children: Nystatin oral suspension is classified as FDA pregnancy risk category C. It's also unknown whether nystatin is excreted in human milk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Mean change in S. Mutans carriage | baseline to 3 months
  Subjects' whole non-stimulated saliva samples will be collected by spitting into a sterilized 50ml centrifuge tube. S. mutans will be isolated using Mitis Salivarius with Bacitracin selective medium (37°C for 48h) and identified by colony morphology. S. mutans carriage following nystatin suspension oral application using the colony forming unit and scoring (1: no detection, 2: 1-10,000 CFU/mL; 3: >10,000 CFU/mL). Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Mean C Albicans carriage | baseline to 3 months
  Subjects' whole non-stimulated saliva samples will be collected by spitting into a sterilized 50ml centrifuge tube. BBLTM CHROMagarTM Candida (BD, Sparks, MD, USA) will be used to isolate C. albicans (37°C for 48h). This medium permits presumptive identification of several clinically important Candida species including C. albicans based on colony color and morphology. C. albicans detection and carriage following nystatin suspension oral application using colony forming unit and scoring (1: no detection, 2: 1-400 CFU/mL; 3: >400 CFU/mL).
Mean change in plaque index | baseline to 3 months
  Dental plaque status will be assessed using the Plaque Index. Each of the four gingival areas of the tooth will be given a score from 0-3. A score of 0 indicates no plaque in the gingival area, a score of 1 indicates the presence of a film of plaque adhering to the free gingival margin, a score of 2 indicates moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and or adjacent tooth, a score of 3 indicates abundance of soft matter within the gingival pocket and or on the gingival margin and adjacent tooth structure. The scores of each tooth surface will be added and divided by the number of teeth examined to obtain the plaque index score. Higher scores indicate worse outcome
Mean change in number of bleeding on probing sites | baseline to 3 months
  Bleeding on probing (BOP) will be evaluated to reflect the periodontal status. With a periodontal probe, the periodontal tissue will be assessed to the bottom of the clinical pocket or sulcus. No extra effort will be made to apply a pressure. If bleeding occurs within 10-15 seconds after probing, the positive mark will be recorded on the form. Interproximal sites for every existing tooth, except the third molars, will be scored both from the buccal and the lingual sides. Due to the different numbers of existing teeth for each subject, the change in numbers of BOP sites will be measured and compared.
Mean change in diversity as measured by the Shannon Index | baseline to 3 months
  We will use established methods to perform the oral microbiome sequencing and related bioinformatics analysis. Genomic DNA from clinical samples will be extracted. The bacterial 16S rRNA V1-V3 hypervariable region and fungal ITS region will be amplified and sequenced on an Illumina MiSeq. Absolute abundance of bacteria and fungi in each sample will be determined by quantitative real-time PCR using 16s and ITS primers, probe and cloned plasmid standards. Sequence reads will be assessed for quality using Quantitative Insights into Microbial Ecology software. USearch will be used to identify specific bacteria/fungi or operational taxonomic units using the GreenGenes and UNITE databases of reference sequences. Bacterial diversity within each sample (alpha diversity) will be computed as the Shannon Index. Equitability assumes a value between 0 and 1 with 1 being complete evenness.
Mean change in diversity as measured by the Bray-Curtis dissimilarity index | baseline to 3 months
  We will use established methods to perform the oral microbiome sequencing and related bioinformatics analysis. Genomic DNA from clinical samples will be extracted. The bacterial 16S rRNA V1-V3 hypervariable region and fungal ITS region will be amplified and sequenced on an Illumina MiSeq. Absolute abundance of bacteria and fungi in each sample will be determined by quantitative real-time PCR using 16s and ITS primers, probe and cloned plasmid standards. Sequence reads will be assessed for quality using Quantitative Insights into Microbial Ecology software. USearch will be used to identify specific bacteria/fungi or operational taxonomic units using the GreenGenes and UNITE databases of reference sequences. Bacterial diversity between samples (beta diversity) will be computed as the Bray-Curtis dissimilarity index. The Bray-Curtis dissimilarity is a number between 0 (the two sites share all the same species) and 1 (they do not share any species).

CONTACTS AND LOCATIONS:
Overall Officials: Jin Xiao, DDS, PhD, Principal Investigator — University of Rochester
Locations (1):
- Eastman Dental Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04550546/ICF_000.pdf